CLINICAL TRIAL: NCT01789242
Title: A Phase I Dose Escalation Study of Carfilzomib in Patients With Previously-Treated Systemic Light-Chain (AL) Amyloidosis
Brief Title: A Safety Study of Carfilzomib in Patients With Previously-Treated Systemic Light Chain Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Criterium, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMyC 11MM02; IST-CAR-545 (Other: Onyx Pharmaceuticals)
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Amyloidosis; Systemic Light Chain Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib (Experimental): All eligible subjects will receive the study intervention of Carfilzomib. Patients with suboptimal hematologic responses (<VGPR after 4 cycles) will have Dexamethasone added to their treatment.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — IV over 30 minutes on Days 1, 2, 8, 9, 15, and 16 every 28 days.
  Other Names: PR-171; Kyprolis
Drug: Dexamethasone — Dexamethasone IV or PO on Days 1, 2, 8, 9, 15, and 16 every 28 days in patients with <VGPR after 4 cycles.
  Other Names: Decadron

SUMMARY:
This is a dose finding study to evaluate the safety and determine the maximum tolerated dose of carfilzomib in patients with previously treated systemic light-chain amyloidosis.

DETAILED DESCRIPTION:
This is a dose finding study to evaluate the safety and determine the maximum tolerated dose of carfilzomib in patients with previously treated systemic light-chain amyloidosis. The study will also explore the efficacy of carfilzomib in both proteasome inhibitor-naive and proteasome inhibitor-exposed patients including hematologic response, organ response, progression free survival, and time to next therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Histologically-proven AL amyloidosis, confirmed by positive Congo red stain with green birefringence on polarized light microscopy with evidence of measurable clonal disease that requires active treatment as defined below:
* Patients must have clonal disease measureable by serum free light chain (FreeliteTM) assay:

  * For the dose-escalation cohort: this is defined as having any elevation in the amyloidogenic (i.e. clonal) light chain with an abnormal free kappa:lambda ratio
  * For the dose expansion cohorts: in addition to the above, there must be a difference between the amyloidogenic (i.e. clonal) and non-amyloidogenic light chain (dFLC) of at least 50mg/L (5mg/dL)
* Relapsed (progressed after prior response) or refractory (failed to achieve at least a partial response) to at least one prior therapy for amyloidosis.

  * Patients that received an autologous stem cell transplant must be at least 3 months post-transplant and recovered from acute transplant-related toxicities.
  * Patients that were unable to tolerate at least 1 cycle of an alkylating agent plus corticosteroid (e.g. melphalan + dexamethasone) or alternative prior regimen because of severe adverse events (e.g. hypersensitivity reaction) may be considered after discussion with the study PI/Medical Monitor.
* Objective, measureable, symptomatic organ involvement, defined as one or more of the following:

  * Kidney: albuminuria ≥ 500 mg/day in a 24-hour urine specimen
  * Heart: presence of mean left ventricular wall thickness on echocardiogram greater than 12 mm in the absence of hypertension or valvular heart disease, or unexplained low voltage (< 0.5 mV) on ECG, or NT-proBNP > 332 ng/L in the absence of impaired renal function [estimated glomerular filtration rate (eGFR) < 45 mL/min]
  * Liver: hepatomegaly on physical exam with elevated alkaline phosphatase > 1.5 x ULN
  * GI Tract: biopsy showing amyloid deposition along with symptoms such as GI bleeding or persistent diarrhea (> 4 loose stools/day) Autonomic or Peripheral Nervous System: defined as orthostasis, symptoms of nausea or dysgeusia, recurrent diarrhea or constipation, abnormal sensory and/or motor findings on neurologic exam, or gastric atony by gastric emptying scan
  * Note: Skin, lymph node, or soft tissue involvement; carpal tunnel syndrome; or bone marrow amyloid as the sole clinical manifestations of amyloidosis are not sufficient for inclusion.
* Amyloid cardiac biomarker stage I or II disease Staging defined by NT-proBNP and troponin T cut-offs of < 332 pg/mL and <0.035 ng/mL, respectively, as thresholds: Stage I, both under threshold; and Stage II, either troponin or NT-proBNP (but not both) over threshold. If troponin T is not available at local institution, troponin I may be used, but threshold is <0.1 ng/mL.23
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Clinical laboratory values as specified within 14 days of treatment:

  * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
  * Hemoglobin ≥8 g/dL [transfusion permitted]
  * Platelet count ≥75.0 x 109/L
  * Total bilirubin ≤ 2 x Upper Limit of Normal (ULN)
  * Alkaline phosphatase ≤ 5 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.5 x ULN
  * CrCl ≥ 30 mL/min as measured by 24-hour urine
  * Screening ANC should be independent of granulocyte-and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for at least 2 weeks
  * Screening platelet count should be independent of platelet transfusions for at least 2 weeks
* Written informed consent in accordance with federal, local, and institutional guidelines
* Females of childbearing potential must agree to ongoing pregnancy testing and to practice contraception or abstain from heterosexual intercourse
* Male patients must agree to practice contraception or to abstain from heterosexual intercourse
* Male patients must agree not to donate semen or sperm
* Life expectancy of ≥ 3 months

Exclusion Criteria:

* Pregnant or lactating females
* Major surgery within 21 days prior to first dose
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 14 days prior to first dose
* Treatment with an experimental drug within 28 days of first dose
* Active Human Immunodeficiency Virus (HIV) or hepatitis B or C infection
* Bone marrow plasma cells ≥ 30% or clinical manifestations of multiple myeloma, such as hypercalcemia or lytic bone lesions
* Cardiac exclusions:

  * Left ventricular ejection fraction (LVEF) < 40%
  * Amyloid cardiac biomarker stage III disease, defined as both NT-proBNP ≥ 332 pg/mL and troponin T ≥ 0.035 ng/mL. If troponin T is not available at local institution, troponin I may be used, but cut-off is ≥ 0.1 ng/mL
  * New York Heart Association (NYHA) classification III or IV heart failure (see Appendix G) despite medical management
  * Unstable angina or myocardial infarction within 6 months prior to first dose
  * Grade 2 or 3 atrioventricular (AV) block (Mobitz type I is permitted) or sick sinus syndrome, unless subject has a pacemaker
  * Known history of sustained (> 30 second) ventricular tachycardia or cardiac syncope. Known history of recurrent non-sustained ventricular tachycardia (> 3 beats) despite anti-arrhythmic therapy
  * Supine systolic blood pressure < 90 mm Hg, or symptomatic orthostatic hypotension, or a decrease in systolic blood pressure upon standing of > 20 mm Hg despite medical management (e.g. midodrine, fludrocortisones)
* Significant peripheral neuropathy (Grade 3, Grade 4, or Grade 2 with pain) within 14 days prior to first dose
* Severe diarrhea (≥ grade 3) not controllable with medication or that requires total parenteral nutrition
* History of bleeding diathesis, known factor X deficiency (level < 20%), or requirement for therapeutic anticoagulation with warfarin
* Known allergies to carfilzomib or Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
* Presence of other active malignancy with the exception of non-melanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate-specific antigen is within normal limits, or any completely resected carcinoma in situ
* Serious psychiatric or medical conditions that could interfere with treatment
* Contraindication to any of the required concomitant drugs, including antiviral (e.g. Valacyclovir)
* Patients in whom the required program of oral and IV fluid hydration is contraindicated, e.g. due to severe pre-existing pulmonary, cardiac, or renal impairment
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events as a Measure of Safety and Tolerability | Throughout treatment, estimated at 8 months per patient
  Review of adverse events for safety and to determine the maximum tolerated dose of the combination treatment

SECONDARY OUTCOMES:
Hematologic Response | Every 28 days while on treatment (estimated at 8 months per patient)
  Hematologic Response Rates (PR, VGPR, and CR
Organ Response | Every 112 days while on treatment (estimated at 8 months per patient)
  Organ response rates by standard criteria
Progression Free Survival | throughout study and follow up (every 2-3 months for 2 years
Time to next therapy | throughout follow up (every 2-3 months for 2 years)

OTHER OUTCOMES:
Impact on hematologic response and toxicity of adding dexamethasone | Every 28 days throughout treatment after dexamethasone is added (estimated at 4 months per patient)
  Impact on hematologic response and toxicity of adding dexamethasone to carfilzomib in patients with suboptimal hematologic responses (defined as <VGPR after 4 cycles)
Biomarkers of carfilzomib sensitivity | Baseline
  Evaluate potential biomarkers of carfilzomib sensitivity in baseline purified bone marrow plasma cells, including proteasomal capacity and in vitro sensitivity to proteasome inhibition.
Prognostic significance of cycle D1 expression | Baseline
  To explore the prognostic significance of cyclin D1 expression in purified bone marrow plasma cells in patients with previously treated AL amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, Principal Investigator — AMyC; Univ of Penn Perelman Center for Advanced Medicine; Brian GM Durie, MD, Principal Investigator — AMyC; Raymond Comenzo, MD, Principal Investigator — AMyC, Tufts University
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Boston University Medical Center, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Sciences University, Portland, Oregon
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania